CLINICAL TRIAL: NCT05581966
Title: Wound Assessment Using Spectral Imaging
Brief Title: Wound Assessment Using Spectral Imaging EU/UK
Acronym: WAUSI EU/UK
Status: Completed | Type: Observational
Sponsor: SpectralMD (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-2022-003
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Diabetes; Diabetic Foot; Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Diabetic Foot Ulcer (DFU) Group: Patients with DFUs undergoing 30 day standard wound care (SWC) therapy as part of their standard of care
  Interventions: Diagnostic Test: DV-SSP Imaging

INTERVENTIONS:
Diagnostic Test: DV-SSP Imaging — DeepView utilizes imaging data from DFUs to aid in health care providers' assessment of wound healing potential. It is intended to be used as an aid to health care providers in the management of DFU wounds and not as a standalone prediction device.

SUMMARY:
During the observational, non-interventional study, at Baseline Study Visit (BSV) subjects will be screened and consented. Eligible subjects will undergo imaging with the DeepView device. Pre- and post-debridement images will be obtained (if debridement performed per SOC), as well as reviewing medical history and physical assessments.

Additional Study Visits (SVs) will be performed when patient returns to the clinic for Routine Clinic Visit for up to 12 weeks or wound closure. During these visits DeepView imaging will occur pre- and post-debridement, and the status of the subject's treatment will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Subject has an ulcer, or a slow healing wound that is full thickness for at least 4 weeks, below the malleolus, in the presence of Diabetes.
* The target ulcer will be the largest ulcer if two or more eligible DFUs are present and will be the only one evaluated in the study.
* The target ulcer is planned to undergo standard wound care (SWC) therapy (See 8.6 Standard Wound Care (SWC) Therapy).
* Subject understands and is willing to participate in the clinical study and can comply with required visits.

Exclusion Criteria:

* Target ulcer is deemed by the investigator to be caused by a medical condition other than diabetes.
* Target ulcer, in the opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a carcinoma of the ulcer.
* Eligible DFU has associated untreated acute osteomyelitis or active infection
* Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids >10mg daily dose), or cytotoxic chemotherapy.
* Subjects on any investigational drug(s) or device(s) within 30 days preceding initial study visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with DFUs undergoing SWC treatment
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Data Collection | 12 weeks
  The purpose of this study is to build a database for development and validation of a machine learning (ML) algorithm for diabetic foot ulcer (DFU) healing assessment using images obtained with the Spectral MD DeepView device.

CONTACTS AND LOCATIONS:
Locations (1):
- Connolly Hospital, Diabetic Day Centre, Abbotstown, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No